CLINICAL TRIAL: NCT06985823
Title: Effects of Rotational Versus Anti-rotational Exercises on Endurance, Balance, and Core Stability in Gym-goer
Brief Title: Rotational Versus Anti-Rotational Exercises on Endurance, Balance, and Core Stability in Gym-goer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0455
Record Dates: First submitted 2025-05-15; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Sports Physical Therapy
Keywords: Balance, Core stability, Endurance, Exercise, Rotational
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rotational exercises (Experimental): 14 participants will be in experimental group A, giving them rotational exercises (Rotational Crunch exercise, Single leg romanian deadlift with rotation, rotational medicine ball throws for six weeks. Measure all values before giving them protocol and after protocol.
  Interventions: Other: Rotational exercises
- Anti-Rotational exercises (Experimental): 14 participants will be in experimental group B, giving them anti-rotational exercises (Quadruped exercise 3 sets of 15 repetition, planks 3 sets of 60 second hold, pallof press 3 sets of 15 repetition) for six weeks. Measure all values before giving them protocol and after protocol.
  Interventions: Other: Anti-Rotational exercises

INTERVENTIONS:
Other: Rotational exercises — 14 participants will be in experimental group A, giving them rotational exercises (Rotational Crunch exercise, Single leg romanian deadlift with rotation, rotational medicine ball throws for six weeks. Measure all values before giving them protocol and after protocol.
  Arms: Rotational exercises
Other: Anti-Rotational exercises — 14 participants will be in experimental group B, giving them anti-rotational exercises (Quadruped exercise 3 sets of 15 repetition, planks 3 sets of 60 second hold, pallof press 3 sets of 15 repetition) for six weeks. Measure all values before giving them protocol and after protocol.
  Arms: Anti-Rotational exercises

SUMMARY:
Core exercises play an important role in improving the overall fitness of gym-goer. They improve core stability, which is essential for maintaining proper posture and reducing the risk of injuries during workouts. Core exercises also help improve balance and coordination, which are important for daily activities and sports. Rotational exercises involve twisting movements that engage the core, while anti-rotational exercises focus on resisting twisting forces to enhance core stability.

It is a randomized clinical trial with non-probability convenience sampling technique. The sample size of the study is 28. It will be conducted in one rep fitness club and 360 fitness club in Lahore within 6 months after approval of synopsis. Participants in group A (Rotational exercise group) attended 3 times per week with 15 repetitions (3 sets of 15 repetitions) and approximately 30-45 minutes per session, for six weeks. Each training program led the participants followed by a series of exercises, (Rotational Crunch exercise, Single leg romanian deadlift with rotation, rotational medicine ball throws). Participants in group B (Anti-Rotational exercise group) attended 3 times per week, approximately 30-45 minutes per session, for six weeks. Training program led the participants followed by a series of exercises, (Quadruped exercise 3 sets of 15 repetition, planks 3 sets of 60 second hold, pallof press 3 sets of 15 repetition). The collected data will be analyzed in Statistical Package for the Social Sciences (SPSS) 25.0. If data will be normally distributed, then parametric; if not normally distributed, then non-parametric.

The aim of the study is to compare the effects of rotational versus anti-rotational exercises on endurance, balance, and core stability in gym-goer.

DETAILED DESCRIPTION:
The objective of my study is to determine comparative effects of rotational versus anti-rotational exercises on endurance, balance, and core stability in gym-goer.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-30 years
* Only female participants
* Females who have been consistently engaging in gym-based exercise for a minimum duration of 6 months up to 1 year

Exclusion Criteria:

* Participants was excluded if they have a leg length discrepancy
* History of serious musculoskeletal injuries or conditions (Fractures, Dislocations) within past 6 months.
* Females who are pregnant (All trimesters) or within the postpartum period
* Systematic conditions: Diabetic, Hypertension

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Females are eligible to participate.
Enrollment: 28 (Actual)
Dates: Start 2024-07-30 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Planks | Time Frame: 6 weeks
  An exercise in which you hold your body straight and parallel to the floor while resting on your toes and hands or elbows. Planks are very good for endurance and strengthening your core.
Star Excursion Balance Test (SEBT) | Time Frame: 6 weeks
  The Star Excursion Balance Test (SEBT) is a dynamic test that requires strength, flexibility, and proprioception. It is a measure of dynamic balance that provides a significant challenge to athletes and physically active individuals.
  The points that are measured: Anterior, Posterior, Medial, Lateral, Anteromedial, Anterolateral, Posteromedial, Posterolateral.
  If the patient uses the right leg to reach, they would follow this in clockwise order. If they use the left leg to reach, they would follow this in anti-clockwise order.
Sahrmann core stability test | Time Frame: 6 weeks
  The Sahrmann five-level core stability test was assumed to evaluate the abdominal muscle function as they act by isometrically contracting into flexion to maintain lumbar spine flexion by posteriorly tilting the pelvis against an assumed increasing resistance.

CONTACTS AND LOCATIONS:
Overall Officials: Aamir Gul Memon, MS, Principal Investigator — Riphah International University
Locations (1):
- 360 Fitness club and One Rep Fitness club, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nakai Y, Kawada M, Miyazaki T, Kiyama R. Trunk muscle activity during trunk stabilizing exercise with isometric hip rotation using electromyography and ultrasound. J Electromyogr Kinesiol. 2019 Dec;49:102357. doi: 10.1016/j.jelekin.2019.102357. Epub 2019 Sep 16. PMID 31557703
- [Background] Zemkova E, Zapletalova L. Back Problems: Pros and Cons of Core Strengthening Exercises as a Part of Athlete Training. Int J Environ Res Public Health. 2021 May 18;18(10):5400. doi: 10.3390/ijerph18105400. PMID 34070164
- [Background] Oliva-Lozano JM, Muyor JM. Core Muscle Activity During Physical Fitness Exercises: A Systematic Review. Int J Environ Res Public Health. 2020 Jun 16;17(12):4306. doi: 10.3390/ijerph17124306. PMID 32560185
- [Background] Cabrejas C, Solana-Tramunt M, Morales J, Nieto A, Bofill A, Carballeira E, Pierantozzi E. The Effects of an Eight-Week Integrated Functional Core and Plyometric Training Program on Young Rhythmic Gymnasts' Explosive Strength. Int J Environ Res Public Health. 2023 Jan 6;20(2):1041. doi: 10.3390/ijerph20021041. PMID 36673798
- [Background] Palmer TG, McCabe M. The Effect of a Novel Weight-Supported Kinetic Chain Resistance Training Program on Proximal Core Muscular Endurance, Trunk-to-Arm Muscular Power, and Bat Swing Speed. J Strength Cond Res. 2023 Nov 1;37(11):2130-2140. doi: 10.1519/JSC.0000000000004520. PMID 37883393
- [Background] Ylinen J, Pasanen T, Heinonen A, Kivisto H, Kautiainen H, Multanen J. Trunk muscle activation of core stabilization exercises in subjects with and without chronic low back pain. J Back Musculoskelet Rehabil. 2024;37(4):897-908. doi: 10.3233/BMR-230043. PMID 38250755
- [Background] Watanabe Y, Kato K, Otoshi K, Tominaga R, Kaga T, Igari T, Sato R, Oi N, Konno SI. Associations between core stability and low back pain in high school baseball players: A cross-sectional study. J Orthop Sci. 2022 Sep;27(5):965-970. doi: 10.1016/j.jos.2021.05.010. Epub 2021 Jun 22. PMID 34167867
- [Background] Powden CJ, Dodds TK, Gabriel EH. THE RELIABILITY OF THE STAR EXCURSION BALANCE TEST AND LOWER QUARTER Y-BALANCE TEST IN HEALTHY ADULTS: A SYSTEMATIC REVIEW. Int J Sports Phys Ther. 2019 Sep;14(5):683-694. PMID 31598406
- [Background] Choi JH, Kim DE, Cynn HS. Comparison of Trunk Muscle Activity Between Traditional Plank Exercise and Plank Exercise With Isometric Contraction of Ankle Muscles in Subjects With Chronic Low Back Pain. J Strength Cond Res. 2021 Sep 1;35(9):2407-2413. doi: 10.1519/JSC.0000000000003188. PMID 31136542
- [Background] Mo RCY, Ngai DCW, Ng CCM, Sin KHS, Luk JTC, Ho IMK. Effects of loading positions on the activation of trunk and hip muscles during flywheel and dumbbell single-leg Romanian deadlift exercises. Front Physiol. 2023 Nov 29;14:1264604. doi: 10.3389/fphys.2023.1264604. eCollection 2023. PMID 38093908